CLINICAL TRIAL: NCT04116320
Title: Pilot Evaluation of Focused Ultrasound Ablation and Focused Ultrasound Ablation Plus PD-1 Antibody Blockade in Advanced Solid Tumors
Brief Title: Focused Ultrasound Ablation and PD-1 Antibody Blockade in Advanced Solid Tumors
Acronym: AM-003
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to enroll enough patients to complete targeted enrollment in a reasonable time.
Sponsor: Craig L Slingluff, Jr (Other)
Collaborators: Theraclion (Industry)
Responsible Party: Sponsor-Investigator, Craig L Slingluff, Jr, Professor of Surgery; Director, Human Immune Therapy Center, University of Virginia
Organization: University of Virginia (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21850
Record Dates: First submitted 2019-10-03; First posted 2019-10-04 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2023-08

CONDITIONS: Melanoma; Breast Cancer; Merkel Cell Carcinoma; Squamous Cell Cancer; Non Small Cell Lung Cancer; Cervical Cancer; Urothelial Carcinoma; Ovarian Cancer; Hepatocellular Carcinoma; Small-cell Lung Cancer; Microsatellite Instability High; Gastric Cancer; Esophageal Cancer
Keywords: Echopulse; Focused Ultrasound Ablation; FUSA; Pembrolizumab; Keytruda; Atezolizumab; Tecentriq; polyICLC; poly-ICLC; Hiltonol
MeSH Terms: conditions — Melanoma; Breast Neoplasms; Carcinoma, Merkel Cell; Neoplasms, Squamous Cell; Carcinoma, Non-Small-Cell Lung; Uterine Cervical Neoplasms; Carcinoma, Transitional Cell; Ovarian Neoplasms; Carcinoma, Hepatocellular; Small Cell Lung Carcinoma; Stomach Neoplasms; Esophageal Neoplasms | interventions — High-Intensity Focused Ultrasound Ablation; poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Cohort 1, primary regimen (Regimen 1a) (Experimental): FUSA therapy and standard of care PD-1 blockade. FUSA therapy will be administered on day 8.
  Interventions: Device: Echopulse; Drug: Standard of Care PD-1 Therapy
- Cohort 1, secondary regimen (Regimen 2a) (Experimental): FUSA therapy, standard of care PD-1 blockade, and intratumoral poly-ICLC will be administered on day 8.
  Interventions: Device: Echopulse; Drug: Poly ICLC; Drug: Standard of Care PD-1 Therapy
- Cohort 2, primary regimen (Regimen 1b) (Experimental): FUSA therapy will be administered on day 1.
  Interventions: Device: Echopulse
- Cohort 2, secondary regimen (Regimen 2b) (Experimental): FUSA therapy and intratumoral poly-ICLC will be administered on day 1.
  Interventions: Device: Echopulse; Drug: Poly ICLC

INTERVENTIONS:
Device: Echopulse — The Echopulse device delivers focused ultrasound ablation (FUSA) therapy. FUSA is a technology that delivers continuous high-intensity focused ultrasound to ablate tissue.
  Other Names: Focused Ultrasound Ablation; FUSA
Drug: Poly ICLC — Poly-ICLC is a TLR3 agonist.
  Other Names: Hiltonol
  Arms: Cohort 1, secondary regimen (Regimen 2a); Cohort 2, secondary regimen (Regimen 2b)
Drug: Standard of Care PD-1 Therapy — PD-1 therapy FDA approved for use on a 3-week schedule will be used per standard of care.
  Arms: Cohort 1, primary regimen (Regimen 1a); Cohort 1, secondary regimen (Regimen 2a)

SUMMARY:
This study evaluates whether it is safe to Focused Ultrasound Ablation (FUSA) treatments with and without PD-1 blockade and with and without intratumoral poly-ICLC. A device called the Echopulse will be used for the FUSA therapy. Patients will be assigned to 1 of 2 cohorts depending on their disease and treatment status. In Cohort 1, patients will receive FUSA therapy while receiving PD-1 blockade therapy as part of standard clinical care treatment. In Cohort 2, patients who discontinue or are ineligible for PD-1 blockade therapy will undergo FUSA without concurrent systemic therapy, with the goal of utilizing the FUSA to boost the innate immune response. The optional secondary regimen will combine FUSA (+/- PD-1 blockade) with intratumoral poly-ICLC.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Advanced solid tumor with measurable disease.
3. Subject must have failed or have contraindication to standard therapies.
4. For Cohort 1, primary regimen (Regimen 1a): Patients with advanced solid malignancy for which PD1 or PDL1 antibody monotherapy administered on a 3-week schedule is FDA-approved for treatment, who have one or more tumor deposits that are accessible to focused ultrasound treatment, and who are eligible to receive (or to continue to receive) PD1 or PDL1 blockade therapy. Uveal melanoma patients are not eligible for Regimen 1a.

   Note: Participants eligible for this regimen may receive the primary protocol therapy (Regimen 1a) concurrent with PD1/PDL1 antibody therapy if:
   * Progressive Disease: subjects with progressive disease following PD1/PDL1 antibody therapy are eligible for this cohort if it is clinically appropriate for them to continue on systemic PD1/PDL1 antibody per the treating clinician even if they did not begin treatment on this trial. Examples may include a patient with a small new lesion but stable disease in other sites, or very slight tumor growth in multiple sites, in a patient without other approved therapy options. Participants who progress following PD1/PDL1 antibody therapy may undergo interval resection of enlarging lesions and still be included in this cohort as long as they have persistent unresectable disease that is accessible to FUSA treatment.
   * Response with persistent disease: subjects who have a clinical response (SD or PR) and have residual lesion(s) accessible to FUSA treatment. Participants with PR are only eligible if it is clinically appropriate for them to continue on PD1/PDL1 therapy per the judgement of the treating clinician.
   * Stable disease: The majority of clinical responses to PD1/PDL1 blockade occur within 12 weeks but may occur much later. Routine clinical practice commonly includes continuation of PD1 antibody therapy for 1-2 years for patients with stable disease on that therapy. Thus, patients with SD after 12 weeks of PD1/PDL1 therapy per RECIST criteria may be eligible for Regimen 1a if their disease has remained stable on therapy and if their treating provider recommends continuation of PD1/PDL1 therapy even if they were not treated on this trial.
5. For Cohort 1, secondary regimen (Regimen 2a): For those patients treated with primary regimen 1a, select participants may be enrolled in a secondary regimen. This would include participants in the following scenarios:

   * Stable disease.
   * Response in lesion treated in regimen 1, but persistent disease or progression in a separate lesion.
   * Initial partial response but still persistent disease at the treated lesion.
   * Initial response followed by progression at treated lesion or separate site, after discontinuation of PD-1/PD-L1 antibody. If there is a response and then progression at the site treated in Regimen 1 and the residual tumor meets inclusion criteria, this lesion may be re-treated on the secondary regimen.
   * Participants with lesions unique from the lesion treated in regimen 1 may enroll in regimen 2 and have additional lesion(s) treated, as long as they meet all inclusion criteria requirements. Up to three lesions may be treated in the second regimen.

   Patients enrolling to Regimen 2a must have a target lesion amenable to intratumoral injection with polyICLC per the treating clinician's discretion. The lesion(s) to be FUSA treated in regimen 2 do not need to include the lesion targeted in regimen 1. The patient must remain eligible for PD1/PDL1 Ab therapy.
6. For Cohort 2, primary regimen (Regimen 1b): The following patient subsets would be eligible for the Cohort 2 primary regimen, as long as they have failed (progressed or not tolerated) or are not eligible for all effective available approved therapies known to confer clinical benefit:

   * Patients with advanced solid malignancy for which PD1 or PDL1 blockade is not FDA-approved.
   * Patients with metastatic uveal melanoma
   * Patients with advanced solid malignancies for which PD1 or PDL1 blockade is FDA approved but who are not eligible to receive that therapy because of prior failure, toxicity, baseline autoimmune disease, or frailty.
   * Patients who previously responded to PD1/PDL1 therapy but then progressed, if there are no other systemic therapies available to them.

   Patients who were previously undergoing PD-1 blockade therapy must not have received a dose within 4 weeks prior to FUSA treatment.
7. For Cohort 2, secondary regimen (Regimen 2b): For those patients treated with primary regimen 1a or 1b, select participants may be enrolled in a secondary regimen. This would include participants in the following scenarios:

   * Stable disease.
   * Response in lesion treated in regimen 1, but persistent disease or progression in a separate lesion.
   * Initial partial response but still persistent disease at the treated lesion.
   * Initial response followed by progression at the treated lesion after discontinuation of PD-1/PD-L1 antibody. If there is a response and then progression at the site treated in Regimen 1 and the residual tumor meets inclusion criteria, this lesion may be re-treated on the secondary regimen. For participants who progress at a site unique from the treated lesion, they may enroll in Regimen 2 and have this new lesion treated, as long as they meet all inclusion criteria requirements.
   * Participants with lesions unique from the lesion treated in regimen 1 may enroll in regimen 2 and have additional lesion(s) treated, as long as they meet all inclusion criteria requirements. Up to three lesions may be treated in the second regimen.

   Patients enrolling to Regimen 2b must have a target lesion amenable to intratumoral injection with polyICLC per the treating clinician's discretion. The lesion to be FUSA treated in regimen 2 does not need to be the same lesion targeted in regimen 1. Crossover from primary regimen 1a is allowed if the patient is no longer eligible for continued PD1/PDL1 Ab therapy (e.g. due to autoimmune toxicity), and if there is no other effective systemic therapy option. The length between the FUSA treatments in regimen 1 and regimen 2 should be no less than 6 weeks. Patients who experienced an unanticipated device effect in the primary regimen are not eligible for the secondary regimen.
8. One or more dermal, subcutaneous or nodal metastases from an advanced solid tumor. The metastases need to be accessible for FUSA and for biopsy.

   For FUSA:

   The targeted lesion(s) must be visible by ultrasound imaging and meet the following criteria. Brain lesions may not be targeted for treatment.
   * Approximately 1 cm (or more) diameter of treatable tumor volume for lesions to be treated with FUSA.
   * The target treatment area needs to be contained within a region at least 5 mm from the skin surface and less than or equal to 23 mm from the skin surface.
   * The target treatment area must be at a safe distance from all critical structures, including but not limited to ribs or other bony structures, vital organs, named blood vessels or nerves.
   * The critical structures, with the exception of the skin, will not be in the pre-focal ultrasound path.
   * The anterior-posterior dimension of the treatment area by US should be no less than 9mm.

   For Biopsies:

   Biopsies may be completed with or without image guidance.
9. Lesions that have been selected for focused ultrasound or lesions that have been selected for biopsies as untreated controls may have been previously radiated provided:

   * The tumor site that was previously radiated has progressed.
   * A baseline biopsy of the tumor site is obtained following progression and prior to study entry.
10. ECOG performance status 0-2.
11. Subjects with brain metastases may participate if all of the following are true:

    * There has been no evident growth of any brain metastasis since the most recent treatment
    * No brain metastasis is > 2 cm in diameter at the time of registration.
    * Neurologic symptoms have returned to baseline,
    * There is no evidence of new or enlarging brain metastases,
    * Subjects are not using steroids for at least 7 days prior to registration. Regardless of dose, however, subjects who are on a steroid taper for management of brain metastases are not eligible until 7 days after completion of that steroid taper.
    * Brain metastases will not be targeted for FUSA treatment.
12. Adequate organ function
13. Ability and willingness to give informed consent.

Exclusion Criteria:

A subject will be excluded from participating in the trial if the subject:

1. Has received the following medications or treatments at any time within 3 weeks of study day 1:

   1. Immune therapies including:

      * interferon (e.g. Intron-A®),
      * checkpoint blockade therapies other than anti-PD-1/PD-L1 antibodies,
      * antibodies to costimulatory molecules (e.g. CD27, CD137),
      * small molecule immune therapies (e.g. IDO1 inhibitor)
   2. Cytotoxic chemotherapy for cancer
2. Has received the following medications or treatments at any time within 4 weeks of study day 1:

   1. Radiation therapy (Note: Stereotactic radiotherapy, such as gamma knife, can be used ≥ 1 week prior to registration)
   2. Allergy desensitization injections
   3. High doses of systemic corticosteroids, with the following qualifications and exceptions:

      * Daily doses of 10 mg or less prednisone (or equivalent) per day administered parenterally or orally are allowed in patients with normal adrenal and pituitary function.
      * In patients with adrenal or pituitary insufficiency replacement steroid doses are allowed.
      * Inhaled steroids (e.g.: Advair®, Flovent®, Azmacort®) are permitted at low doses (less than 500 mcg fluticasone per day, or equivalent)
      * Topical and nasal corticosteroids are acceptable.
   4. Growth factors (e.g. Procrit®, Aranesp®, Neulasta®)
   5. Interleukins (e.g. Proleukin®)
   6. Any investigational therapeutic agent (participation in the UVA AM004 clinical trial is permitted)
   7. Targeted therapies specific for mutated BRAF or for MEK
   8. Live vaccine
3. Has a known addiction to alcohol or drugs and is actively taking those agents, or has recently (within 1 year) taken these agents or has ongoing illicit IV drug use.
4. Is HIV positive or has evidence of active Hepatitis B or C virus with some exceptions.
5. Is currently receiving nitrosoureas or has received this therapy within the preceding 6 weeks
6. Is pregnant or breastfeeding. Female participants of childbearing potential must have a negative pregnancy test obtained within 2 weeks prior to registration. Males and females must agree, in the consent form, to use effective birth control methods during the course of treatment and following treatment in accordance with the labeling guidelines for each approved therapy.
7. Has a medical contraindication or potential problem in complying with the requirements of the protocol in the opinion of the investigator.
8. Has an active infection requiring systemic therapy.
9. Has Class III or IV heart disease as classified according to the New York Heart Association.
10. Has had prior autoimmune disorders requiring cytotoxic or immunosuppressive therapy,or autoimmune disorders with visceral involvement. Participants with an active autoimmune disorder requiring these therapies are also excluded.

    Note: The following are not exclusionary:
    * The presence of laboratory evidence of autoimmune disease (e.g. positive ANA titer) without symptoms
    * Clinical evidence of vitiligo
    * Other forms of depigmenting illness
    * Mild arthritis requiring NSAID medications
    * A history of immune-related adverse events with immune therapy, if the immune-related adverse events have resolved to grade 1 or lower.
11. History of another cancer

    Note: the following diagnoses are exceptions and are permitted as long as they have been treated successfully and without clinical evidence of disease:
    * Any cancer that has been treated successfully, without evidence of subsequent recurrence or metastasis for over 5 years
    * Any cancer without distant metastasis that has been treated successfully, without evidence of recurrence or metastasis for over 2 years
    * Squamous cell cancer of the skin without known metastasis
    * Basal cell cancer of the skin without known metastasis
    * Carcinoma in situ of the breast (DCIS or LCIS)
    * Carcinoma in situ of the cervix
12. 12) Previous treatment with polyICLC within 4 weeks. If a subject was previously treated with intratumoral polyICLC and experienced a significant (grade ≥3) toxicity related to the polyICLC treatment, the tumor that was treated should not be re-treated as part of this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
To assess the safety and toxicity of FUSA administered alone or in combination with PD-1 antibody blockade. | 30 days after the last study intervention
  Incidence and severity of adverse events and incidence of dose-limiting toxicities (DLTs).
To estimate the proportion of patients with increased CD8+ T cell infiltration of spot FUSA-treated metastasis. | Day 43 (cohort 1) or Day 36 (cohort 2)
  Proportion of participants achieving at least a 2-fold increase in CD8+ T cell infiltration per mm2.

SECONDARY OUTCOMES:
To estimate the proportion of patients with increased CD8+ T cell infiltration, after spot FUSA, in untreated metastasis, when available. | Day 43 (cohort 1) or Day 36 (cohort 2)
  Proportion of participants achieving at least a 2-fold increase in CD8+ T cell infiltration per mm2

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Dengel, MD, MSc, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results of this study may be shared.
Supporting Information: Study Protocol
Time Frame: Data may be available after the main findings from the final research data set have been accepted for publication.
Access Criteria: Requests for data access will be accepted only with an accompanying signed Data Access Agreement.

REFERENCES:
- [Derived] Sheybani ND, Witter AR, Thim EA, Yagita H, Bullock TNJ, Price RJ. Combination of thermally ablative focused ultrasound with gemcitabine controls breast cancer via adaptive immunity. J Immunother Cancer. 2020 Aug;8(2):e001008. doi: 10.1136/jitc-2020-001008. PMID 32819975